CLINICAL TRIAL: NCT00311259
Title: Melatonin Treatment and Inflammation, Oxidative Stress and Autonomic Function in Connection With Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Other Study IDs: 2612-3108
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2006-04-05 (Estimated); Status verified 2006-02

CONDITIONS: Oxidative Stress; Inflammatory Stress; Myocardial Ischaemia
MeSH Terms: conditions — Coronary Artery Disease | interventions — Melatonin; Pharmaceutical Preparations

STUDY DESIGN:
Time Perspective: Other

INTERVENTIONS:
Drug: Melatonin (drug)
Drug: Laktose

SUMMARY:
The purpose of this study is to determine whether treatment with melatonin can reduce cell damage and inflammation in connection with laparoscopic gall bladder surgery.

DETAILED DESCRIPTION:
Laparoscopic gall bladder surgery is connected with changes in the body resulting in cell damage and inflammation. Melatonin is a hormone produced in brain and regulate sleep rhythm, temperature, production of other hormones and function of organs. Furthermore melatonin can modify cell damage and inflammation. After surgery the production of melatonin is disturbed. The purpose of this study is therefore to determine whether treatment with melatonin can reduce cell damage and inflammation in connection with laparoscopic gall bladder surgery.

ELIGIBILITY:
Inclusion Criteria:

* indikation for laparoscopic cholecystectomy
* women between 18 and 70 years old

Exclusion Criteria:

* men
* acute cholecystectomy
* pancreatitis
* renal insufficient
* well-known liver insufficient
* cardiovascular disease (arrhythmia, well-known ischaemic heart disease)
* drug therapy (digoxin, Ca-antagonist, amiodaron, beta-blocker)
* anticoagulation therapy (marevan and marcoumar)
* praeoperative therapy with opioid, anxiolytica and hypnotica)
* well-known sleep disease
* endocrine disease in drug therapy (diabetes mellitus, thyroid disease)
* daily alcohol consumption (more than 5 drinks)
* bad compliance (language difficulty, mental problems etc.)
* pregnancy and breast-feeding
* lack of written consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-05; Study Completion 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Bülent Kücükakin, Principal Investigator — Department of Surgical Gastroenterology, University Hospital of Copenhagen in Gentofte
Locations (1):
- Department of Surgical Gastroenterology, University Hospital of Copenhagen in Gentofte, Hellerup, Denmark

REFERENCES:
- [Derived] Kucukakin B, Klein M, Lykkesfeldt J, Reiter RJ, Rosenberg J, Gogenur I. No effect of melatonin on oxidative stress after laparoscopic cholecystectomy: a randomized placebo-controlled trial. Acta Anaesthesiol Scand. 2010 Oct;54(9):1121-7. doi: 10.1111/j.1399-6576.2010.02294.x. PMID 20887414